CLINICAL TRIAL: NCT02294877
Title: A Multicenter, Multinational, Observational Morquio A Registry Study (MARS)
Acronym: MARS
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: 110-504
Record Dates: First submitted 2014-10-28; First posted 2014-11-19 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Mucopolysaccharidosis IV Type A; Morquio A Syndrome; MPS IVA
MeSH Terms: conditions — Mucopolysaccharidosis IV | interventions — GALNS protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Blood serum; urine samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vimizim® (elosulfase alfa) — Recombinant human N acetylgalactosamine 6 sulfatase (rhGALNS)
  Other Names: BMN 110

SUMMARY:
The objectives of this program are: to characterize and describe the Mucopolysaccharidosis IV type A (MPS IVA) population as a whole, including the heterogeneity, progression, and natural history of MPS IVA; to evaluate the long-term effectiveness and safety of Vimizim®, including, but not limited to, the occurrence of serious hypersensitivity reactions, anaphylaxis, and changes in antibody status; to help the medical community with the development of recommendations for monitoring MPS IVA patients and reports on patient outcomes to optimize patient care; to collect data on other treatment paradigms, and evaluate the prevalences of their use and their effectiveness; to characterize the effects and safety of Vimizim treatment 5 years from enrollment in the Registry for patients under 5 years of age; to monitor pregnancy exposure, including maternal, neonatal, and infant outcomes; and to monitor patients who have completed the MOR-005 and MOR-007 clinical trials. These patients will be encouraged to enroll in the applicable Registry Substudy and will be monitored using the MOR-005 and MOR-007 assessment schedules, respectively.

DETAILED DESCRIPTION:
MARS is a multicenter, multinational, observational disease registry for patients diagnosed with Mucopolysaccharidosis Type IVA (MPS IVA). The Registry will collect medical history, and clinical and safety assessments every six months, for up to 10 years. The Registry will enroll and collect data on patients over a period of at least 8 years from the time of the first marketing approval globally and data on individual patients will continue to be collected for at least 2 years from the time the last patient was enrolled or until the Registry is completed.

These assessments are designed to further characterize the spectrum of clinical signs and symptoms of the disease, and to further characterize the safety profile of Vimizim in a broader population. It is not required that patients receive Vimizim to be eligible to participate in this Registry.

In addition, this Registry will collect additional data on patients who have completed the MOR-005 and MOR-007 clinical trials. The MOR-005 and MOR-007 clinical trial patients will be enrolled into the appropriate Registry Substudy for a minimum of 5 years from the time of the patient's enrollment in the MOR-005 clinical study or MOR-007 clinical study. After the 5 year period, these patients should remain in MARS until the Registry is complete.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible to participate in this Registry must meet all of the following criteria:

* Diagnosed with MPS IVA as confirmed by either N-acetylgalactosamine 6-sulfatase (GALNS) enzymatic test or by a diagnostic molecular test
* Willing and able to provide written, signed informed consent, or, in the case of patients age < 18 years, provide written assent (if required) and written informed consent, signed by a legally authorized representative after the nature of the Registry has been explained and prior to performance of any Registry-related procedures
* Willing to undergo assessments to establish baseline data or permit Investigator to enter assessment data recorded prior to Registry entry if available in the patient's medical records. Entry assessments may include: demographics, medical history, urinary keratan sulfate level, urinary protein level, immunogenicity testing, vital signs, physical examination, and height and weight

Patients eligible to participate in the Registry Substudy for MOR-005 must meet all of the following criteria:

* Must have completed the MOR-005 clinical trial
* Willing and able to provide written, signed informed consent, or, in the case of patients age < 18 years, provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the Registry Substudy has been explained and prior to any Registry-related Substudy procedures
* Willing to permit Investigator to enter assessment data recorded prior to Registry
* Substudy entry if available in the patient's medical records

Patients eligible to participate in this Registry Substudy for MOR-007 must meet all of the following criteria:

* Must have completed the MOR-007 clinical trial
* Willing and able to provide written, signed informed consent, or in the case of patients age < 18 years, provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the Registry Substudy has been explained, and prior to any Registry-related Substudy procedures
* Willing to permit Investigator to enter assessment data recorded prior to Registry Substudy entry if available in the patient's medical records

Exclusion Criteria:

Patients who meet the following exclusion criterion will not be eligible to participate in the Registry or Registry Substudies:

• Patients currently participating in a BMN 110 (elosulfase alfa) clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with MPS IVA disease and patients treated with Vimizim, although patients are not required to receive Vimizim to be eligible to participate in this Registry.
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2014-09; Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Safety of Vimizim treated patients as measured by the incidences of Adverse Events, Serious Adverse Events, and immunology tests | 10 Years
  Additional safety measures are medications, occurrence of Bone Marrow Transplant/Hematopoietic Stem Cell Transplant, clinical laboratory tests, vital signs, Electrocardiograms, Echocardiograms, immunogenicity results, physical examinations, imaging studies, and cervical spine imaging.
  All assessments in this observational study will be carried out per the participating institution's standard of care.
  The MARS Annual report will descriptively summarize the safety and outcome measurements for the duration of this voluntary, observational study.
Efficacy of Vimizim as measured by the 6MWT, 3MSCT, RFTs, FEV1, FIVC, FVC, and MVV | 10 years
  Efficacy of Vimizim as measured by the changes in the 6 minute walk test (6MWT), 3 minute stir climb test (3MSCT), respiratory function tests (RFTs) including forced expiratory volume for 1 second (FEV1), forced inspiratory vital capacity (FIVC), forced vital capacity (FVC), and maximum voluntary ventilation (MVV) and by urinary Keratan Sulfate.

SECONDARY OUTCOMES:
The MARS Pregnancy Substudy will collect safety data measured by Adverse Events, Serious Adverse Events, immunology tests, and the infant outcomes as measured by a live birth | 10 years
  The MARS Pregnancy Substudy will collect safety data on the outcomes of pregnancy in women who receive Vimizim as measured by Adverse Events, Serious Adverse Events, immunology tests, and the infant outcomes as measured by a live birth.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (79):
- United States (26):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - A.I. Dupont Hospital for Children, Wilmington, Delaware
  - Children's National Health System, Washington D.C., District of Columbia
  - Miami Children's Hospital, Miami, Florida
  - Emory University, Decatur, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - University Of Iowa, Iowa City, Iowa
  - University of Louisville Research Foundation Inc. - Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Children's Hospital of Boston, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Specialty Center of Nevada, Las Vegas, Nevada
  - Atlantic Health System, Morristown, New Jersey
  - NYU-Langone Medical Center School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - UTHealth McGovern Medical School, Houston, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (7):
  - Perth Children's Hospital, Perth, Nedlands
  - Children's Hospital of Westmead, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Children's Health Queensland Hospital and Health Service, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Children's Hospital - Victoria, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Austria (2):
  - Universitätsklinik Graz, Graz
  - Medical University of Vienna, Vienna
- Antwerp University Hospital, Edegem, Belgium
- Canada (5):
  - Adult Metabolic Diseases Clinic Vancouver General Hospital, Vancouver, British Columbia
  - Children's & Women's Centre of British Columbia, Vancouver, British Columbia
  - Sainte-Justine Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
- Klinika Dětského a Dorostového Lékařstvi, Prague, Czechia
- Copenhagen University Hospital, Klinik For Sjaeldne Handicap, Copenhagen, Dk-2100, Denmark
- France (3):
  - Hôpital Femme Mère Enfant, Bron
  - Hospital Necker, Paris
  - Hopital d'enfants - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Temple Street Children's University Hospital, Dublin, Ireland
- Italy (4):
  - Azienda Policlinico Vittorio Emanuele, presidio G Rodolico, Università di Catania, Catania
  - Azienda Ospedaliero Meyer, Florence
  - Azienda Ospedaliero San Gerardo di Monza, Monza
  - Federico II University Hospital, Naples
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University of Malay Medical Center, Kuala Lumpur
- Netherlands (2):
  - Academic Medical Center - University of Amsterdam, Amsterdam
  - Rotterdam University Hospital Medical Centre, Rotterdam
- The Children Memorial Health Institute, Warsaw, Poland
- Portugal (3):
  - Hospital Pediátrico de Coimbra (Centro Hospitalar de Coimbra), Coimbra
  - Centro Hospitalar Lisboa Centro - Hospital de Dona Estefânia, Lisbon
  - Centro Hospitalar Lisboa Norte, Lisbon
- San Jorge Children's Hospital, Centro de Investigaciones Clinicas, San Juan, Commonwealth, Puerto Rico
- Taiwan (11):
  - Changhua Christian Hospital (CCH), Changhua, Changhua County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, San-Min District
  - Chang Gung Memorial Hospital, Taoyuan, Taoyuan County
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung Branch, Kaohsiung City
  - China Medical University and Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University (NCKU) Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (8):
  - Belfast City Hospital, Belfast
  - University Hospital Birmingham - Selly Oaks, Birmingham
  - Birmingham Children's Hospital, Birmingham
  - Royal Free NHS Foundation Trust, London
  - National Hospital for Neurology and Neurosurgery, London
  - Great Ormond Street Hospital NHS Foundation Trust, London
  - Royal Manchester Children's Hospital - Manchester University NHS Foundation Trust, Manchester
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No